CLINICAL TRIAL: NCT02215525
Title: Treatment of Chronic HCV Infected Egyptian Patients With Electromagnetic Waves and Herbal Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Egyptian Military Medical Services (Other Government)
Collaborators: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMMS 2014 1
Record Dates: First submitted 2014-06-24; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-07

CONDITIONS: Hepatitis C
Keywords: HCV; UVA; Herbal therapy
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UVA and Herbal (Experimental): Twenty four daily one hour sessions using Extra-corporeal electro-magnetic irradiation device combined with Herbal Food Supplement Selenium containing tables as an Anti Oxidant (Tablet A) starting 10 days before the radiation sessions and to continue for 24 weeks
  Interventions: Device: UVA
- Herbal (Experimental): Chronic HCV patients, non complicated will be treated by Herbal tablets only . 500 mg twice tablets every 6 hours daily for 6 months.
  Interventions: Dietary Supplement: Herbal

INTERVENTIONS:
Device: UVA — device uses UVA
  Other Names: UVA device
  Arms: UVA and Herbal
Dietary Supplement: Herbal — Herbal tablets, 1000 mg every 6 hours daily for 6 months
  Other Names: Herbal tablets
  Arms: Herbal

SUMMARY:
A Randomized, Open-Label, Study to evaluate and compare the efficacy and safety, of extracorporeal irradiation of circulating blood by UVA with antioxidant as a supplement (Selenium containing food supplement herbal tablets) in the treatment of non-cirrhotic subjects with chronic hepatitis C.

DETAILED DESCRIPTION:
Objectives: To evaluate and compare the Efficacy and Safety, of extra-corporeal irradiation of circulating blood by extra-corporeal electro-magnetic irradiation with Selenium containing food supplement herbal tablets in the treatment of non-cirrhotic subjects with chronic hepatitis C.

Background and Rationale: As many as 150 million persons are chronically infected with the hepatitis C virus (HCV) worldwide, and more than 350,000 die annually from liver disease caused by HCV

Egypt is confronted with an HCV disease burden of historical proportions that distinguishes this nation from others. It has the highest prevalence of hepatitis C virus (HCV) in the world, estimated nationally at 14.7% . Approximately, there are 10 million Egyptians carry the virus. Due to its chronic debilitating nature, it has tremendous social and financial impacts on our community. Hence, this trial aims to find a logic rational and effective treatment for Hepatitis C.

Extra-corporeal electro-magnetic irradiation: The wavelength of UV irradiation (UVI) lies in the range of 100-400 nm, and is further subdivided into UVA (315-400 nm), UVB (280-315 nm), and UVC (100-280 nm).UVC and UVB are directly absorbed by DNA bases causing serious DNA damages. On the other hand, DNA damage by UVA is indirect through the formation of Reactive Oxygen Species (ROS) that are formed when other cellular chromophores act as endogenous photo sensitizers. ROS can then react with and damage DNA, or interact with other cell structures such as membranes (lipids) and proteins. All of these different types of damage may hamper cell metabolic processes, such as protein synthesis and cell cycle progression, or induce mutations and cell death . Both Selenium itself and various selenoproteins are proposed to have antioxidant effects, reducing the biological impact of ROS on human cells .

Ultraviolet blood irradiation (UBI) was first used on humans in the early 1930s. The effectiveness of UBI in treating infections was studied extensively in the 1940s and it was found that UBI was extremely successful in treating such infections as peritonitis, pyelitis, sinusitis, puerperal sepsis and wound infections in all but the most advanced cases.Later studies showed UBI helped a number of patients with acute viral hepatitis .Recently, Energex Systems, a developer of advanced UBI technology, studied the effects of UBI therapy on viral loads in 13 patients with the infection and it showed some effect.

Optical and physical characteristics of electro-magnetic irradiation is the narrow band of ultraviolet A radiation with a peak at 365 nm with an average power about 18 µW/cm2 during the session.

For irradiation in the UVA region (315 nm- 400nm) the measured average irradiance was 0.12 mW/cm2in the place of circulating blood at any time of each session(40 sec).

The time integral of irradiance (prescribed exposure dose) is 0.144 J/cm2(1440 J/m2)for total radiant exposure time of 1200 sec (20 min) in all therapeutic sessions (up to maximum of 30 sessions in some particular cases).

The Irradiance power at all bands of output wavelength (250 nm - 1050 nm) from the optical lamps:

Wavelength (nm) Irradiance Power (mW/cm2) Ultraviolet Region A: UVA (315 nm -400 nm) 0.12 mW/cm2 Visible Band: VIS (400 nm - 700 nm) 110.8mW/cm2 Infrared Band: IR (700 nm - 1050 nm) 28.3mW/cm2

Selenium containing herbal food supplement:

No. Name Action

1. Ginseng Liver tonic
2. Saffron Anti - Oxidant
3. Dandelion Anti - Bacterial
4. Curcuma Anti - Parasitic
5. Vinca Rose Anti - Bacterial
6. Wormwood Anti - Oxidant
7. Lemon balm Anti - Bacterial
8. Papay Anti - viral
9. Achillia Anti - viral
10. Arctium Anti - viral
11. Aloe Anti - viral Anti - bacterial Anti - Fungal
12. Asfour Liver support

Detailed Description A Randomized, Open-Label, Study to investigate the Efficacy and Safety of extra-corporeal irradiation of circulating blood with and Selenium containing herbal food supplement tablets in the treatment of non-cirrhotic chronic hepatitis C subjects.

The null hypothesis: There is no difference in outcomes and cure rate of patients with Hepatitis C when using electromagnetic device or herbal tablets containing selenium are used with aim of treatment.

This study was submitted for ethical approval via the relevant Minister of health and Medical military sector Research Ethics Approval Committees.

Study Arm (s)

Interventions (arm 1):

Twenty four daily one hour sessions using Extra-corporeal electro-magnetic irradiation device combined with Herbal Food Supplement Selenium containing tables as an Anti Oxidant (Tablet A) starting 10 days before the radiation sessions and to continue for 24 weeks.

Intervention (arm 2):

Daily Herbal Food Supplement Selenium containing tablets for 24 weeks. What will happen to patients?

1. Invitation to participate:

   Patients with hepatitis C virus infection will be identified from the attendee of the hepatology and tropical diseases clinics at our institute.
2. First Contact:

   Each patient will then receive a phone call from the Research Nurse, to request an indication of whether they would like to participate in the study. If the patient would like to meet face-to-face, in which case arrangement would be made during the investigation tests or outpatient clinic appointments. Otherwise, questions will be answered over the telephone. This phone call is anticipated to last 10 minutes on average.
3. Initial Assessment Meeting and Informed Consent:

   An initial meeting will then take place at which patients will be asked to give their informed consent.

   In addition, demographics, past medical history and baseline observations will be noted. Up-to-date base line investigations will be performed including: FBC, renal functions, liver profile, Viral load PCR. The patients will then be informed of which group they have been randomized into (electromagnetic or herbal tablets). Patients in each group will have a detailed explanation of their corresponding management and booklet will be given to patients to take home.
4. The Electromagnetic Device group:

   Those participants in the intervention group will be invited to attend the treatment cubicles to see the device. They will receive 20 minutes presentation about the theory of the device and how it functions.
5. Repeated Assessment Meetings:

   * The Assessments performed in 3 above, will be repeated:
   * On discharge (-24hrs to +48hrs) with additional returning to normal activities questions.
   * 4-week out-patient appointment in research team clinic.
   * 8-week out-patient appointment in research team clinic
   * 12-week out-patient appointment in research team clinic.
   * 24-week out-patient appointment in research team clinic.
6. Monitoring and Supportive Meetings:

   • The research nurse will be available on the study mobile phone which will be supported by other members of the research team during periods of leave.
7. End of the study:

A final assessment meeting will take place six month after completion of treatment. Participants will be discharged back to the hepatology clinic for long term management. Research team will be notified of any long term adverse effects of either treatment arms.

Last follow up date: 48 weeks from baseline. Recruitment Status: Currently recruiting.

Supervision:

1. The Management and Monitoring Group (MMG). The study will be managed by a 'Management and Monitoring Group' (MMG) which will meet regularly, throughout the study, to manage it and to monitor progress. A Gantt chart showing the points at which MMG meetings are proposed is provided within the appendices. The study management will also comprise 5 sub-groups (involving specialized experts) who will interact with the MMG. A schematic showing all of these study management groups is given in the appendices of this document.

   The MMG will comprise:
   * Patient Representative.
   * Professor Doctor: Tayseer Abdulaal, M.D., Internal medicine, Clinical Immunology Consultant, Egyptian Military Armed Forces
   * Professor Doctor: Mostafa El-Awady, M.D.,Molecular Biology Consultant, Egyptian National Research Center
   * Professor Doctor: Mostafa El-Nakib, M.D., Virology Consultant, Egyptian Military Armed Forces
   * Professor Doctor: Hala Zayed, M.D., Internal medicine, Clinical Immunology Consultant, Egyptian Ministry of Health
   * Professor Doctor: Ahmed El-Sawy, M.D., Gastroenterology Consultant, Egyptian Military Armed ForcesDr
2. The Patient Experience Sub-group The principal sub-group of the MMG will be one who will take responsibility for managing and monitoring the experiences of all patients during the study. This group will comprise Dr Tayseer Abdulaal and the Research Nurses and the Administrator. Therefore, it will be based within the hospital. This group will also be responsible for patient recruitment and for patient data entry onto an appropriate database. This group will make a significant contribution to the overall management of the study (which is done by the MMG) by raising awareness, within that group, of issues relating to all aspects of patient experience that arise as the study progresses.
3. The Critical side effects Sub-group A team of researchers, based at Egyptian military hospital, Ain Shams and Cairo University hospitals will meet within 24 hours of admission of any patients involved in the trial to any of the designated hospital. An action plan will include a thorough evaluation of the patient condition. Ife there is any concern regarding patient safety; the trial will be suspended for further assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the age of 21 and 60 years.
2. Female subjects of childbearing potential must be willing to use effective form of birth control.
3. Sexually active fertile females in childbearing period must have negative results for pregnancy tests.
4. Sexually active fertile males must agree either him or his wife to practicing effective form of birth control.
5. Subject should be treatment: Non cirrhotic HCV chronic Hepatitis.
6. Subjects must be able to understand and to adhere to the study visits schedule.
7. Body mass index (BMI) is >18 to <35kg/m2.
8. Must voluntarily sign and date an informed consent, approved by an Institutional Review Board/Ethics Committee (IRB/EC), prior to the initiation of any study-specific procedures.
9. Chronic HCV for at least 6 months prior to study enrolment. Chronic HCV infection is defined as one of the following:

   * Positive for anti-HCV antibody or HCV RNA at least 6 months before Screening, and positive for HCV RNA and anti-HCV antibody at the time of Screening; OR
   * Positive for anti-HCV antibody and HCV RNA at the time of Screening with a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed prior to enrolment with evidence of chronic hepatitis C disease).
10. Absence of cirrhosis judged by documented results of :-

    * Liver Ultrasound. OR
    * Fibro Test score of ≤ 0.75 and Aspartate Amino transferase to Platelet Ratio Index (APRI) ((AST/AST ULN)X100)/Plt in thousands) ≤ 2 at Screening, OR
    * FibroScan® result of <14.5kPa, OR
    * The absence of cirrhosis based on a liver biopsy within the last 36months.
11. If the rewire multiple assessments on the same date for a subject, fibrosis score was calculated in the order of liver biopsy, FibroScan, and Fibro Test. If the rewire assessments on different dates for a subject by different methods, fibrosis score was calculated n the order of liver biopsy, FibroScan, and Fibro Test. If the rewire assessments on different dates for a subject by the same method, fibrosis score was calculated by maximum value.
12. Subject has a plasma HCV RNA level >10,000 International Units (IU)/mLat screening.

Exclusion Criteria:

1. History of severe, life-threatening or other significant sensitivity to any drug.
2. Females who are pregnant or breast feeding.
3. Recent (within 6-months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol.
4. Positive test result for hepatitis B surface antigen (HbsAg) or anti-HIV antibodies (anti-HIV Ab).
5. Clinically significant abnormalities, other than HCV infection, based upon the results of a medical history, physical examination, vital signs, laboratory profile, a 12-lead electrocardiogram (ECG) and echocardiography that make the subject an unsuitable candidate for this study in the opinion of the Investigator.
6. History of uncontrolled seizures, cancer, or uncontrolled diabetes, as defined by a HbA1C level >8.0%.
7. Any current or past clinical evidence of cirrhosis , a history or presence of ascites, oesophageal varices, or hepatic encephalopathy.
8. Known cause of liver disease other than chronic HCV infection.
9. Screening laboratory analyses show any of the following abnormal laboratory results:

   * Alanine amino transferase (ALT) >5X upper limit of normal (ULN),
   * Aspartate amino transferase (AST) >5X upper limit of normal (ULN),
   * Calculated creatinine clearance (using Cockcroft-Gault method) <50mL/min,
   * Albumin<lower limit of normal (LLN),
   * Prothrombin time INR > 1.5,
   * Haemoglobin < 11 %,
   * Platelets<120,000cellsper mm3
   * Absolute neutrophil count <1500cells/µL,
   * Total bilirubin> 1.5 mg/dL,
10. Clinically significant abnormal echocardiography or ECG.
11. Any contraindications to central venous catheter insertion.
12. Previous history of photosensitivity, skin cancer or presence of a positive family history of Skin Cancer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-10 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
sustained virological response (SVR) at 12 weeks | 12 weeks after the end of treatment
  SVR is defined as an absence of detectable HCV RNA in the serum with use of an assay with a sensitivity of at least 50 IU/mL.

SECONDARY OUTCOMES:
Sustained Virological Response (SVR) at 24 weeks | 24 weeks after completion of the course of treatment.
  Absence of detectable HCV RNA in the serum with use of an assay with a sensitivity of at least 50 IU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Tayseer A Abdulaal, M.D., Principal Investigator — EMMS
Locations (1):
- EMMS, Cairo, Heliopolis, Egypt

REFERENCES:
- [Background] Lindsay KL. Introduction to therapy of hepatitis C. Hepatology. 2002 Nov;36(5 Suppl 1):S114-20. doi: 10.1053/jhep.2002.36226. PMID 12407584
- [Background] Ghany MG, Strader DB, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C: an update. Hepatology. 2009 Apr;49(4):1335-74. doi: 10.1002/hep.22759. No abstract available. PMID 19330875
- [Background] Zeuzem S, Heathcote EJ, Shiffman ML, Wright TL, Bain VG, Sherman M, Feinman SV, Fried MW, Rasenack J, Sarrazin C, Jensen DM, Lin A, Hoffman JH, Sedarati F. Twelve weeks of follow-up is sufficient for the determination of sustained virologic response in patients treated with interferon alpha for chronic hepatitis C. J Hepatol. 2003 Jul;39(1):106-11. doi: 10.1016/s0168-8278(03)00187-9. PMID 12821051
- [Background] Martinot-Peignoux M, Stern C, Maylin S, Ripault MP, Boyer N, Leclere L, Castelnau C, Giuily N, El Ray A, Cardoso AC, Moucari R, Asselah T, Marcellin P. Twelve weeks posttreatment follow-up is as relevant as 24 weeks to determine the sustained virologic response in patients with hepatitis C virus receiving pegylated interferon and ribavirin. Hepatology. 2010 Apr;51(4):1122-6. doi: 10.1002/hep.23444. PMID 20069649
- [Background] Mohamoud YA, Mumtaz GR, Riome S, Miller D, Abu-Raddad LJ. The epidemiology of hepatitis C virus in Egypt: a systematic review and data synthesis. BMC Infect Dis. 2013 Jun 24;13:288. doi: 10.1186/1471-2334-13-288. PMID 23799878
- [Background] Moysan A, Marquis I, Gaboriau F, Santus R, Dubertret L, Morliere P. Ultraviolet A-induced lipid peroxidation and antioxidant defense systems in cultured human skin fibroblasts. J Invest Dermatol. 1993 May;100(5):692-8. doi: 10.1111/1523-1747.ep12472352. PMID 8491992
- [Background] Ridley AJ, Whiteside JR, McMillan TJ, Allinson SL. Cellular and sub-cellular responses to UVA in relation to carcinogenesis. Int J Radiat Biol. 2009 Mar;85(3):177-95. doi: 10.1080/09553000902740150. PMID 19296341
- [Background] Girard PM, Pozzebon M, Delacote F, Douki T, Smirnova V, Sage E. Inhibition of S-phase progression triggered by UVA-induced ROS does not require a functional DNA damage checkpoint response in mammalian cells. DNA Repair (Amst). 2008 Sep 1;7(9):1500-16. doi: 10.1016/j.dnarep.2008.05.004. Epub 2008 Jul 7. PMID 18603484
- [Background] Ferguson LR, Karunasinghe N, Zhu S, Wang AH. Selenium and its' role in the maintenance of genomic stability. Mutat Res. 2012 May 1;733(1-2):100-10. doi: 10.1016/j.mrfmmm.2011.12.011. Epub 2012 Jan 5. PMID 22234051
- [Background] MILEY G, CHRISTENSEN JA. Ultraviolet blood irradiation therapy; further studies in acute infections. Am J Surg. 1947 Apr;73(4):486-93. doi: 10.1016/0002-9610(47)90330-9. No abstract available. PMID 20290583
- [Background] Efficacy of ultraviolet blood irradiation therapy in the control of staphylococcemias. The American Journal of Surgery, Volume 64, Issue 3, June 1944, Pages 313-322
- [Background] OLNEY RC. Treatment of viral hepatitis with the Knott technic of blood irradiation. Am J Surg. 1955 Sep;90(3):402-9. doi: 10.1016/0002-9610(55)90777-7. No abstract available. PMID 13238699
- [Background] George Miley Ultraviolet blood irradiation therapy (Knott technic) in acute pyogenic infections. The American Journal of Surgery, Volume 57, Issue 3, September 1942, Pages 493-50
- See also: New Technology and Methods to Fight Hepatitis C. Nicole Cutler L.Ac. August 6, 2007. — http://www.hepatitiscentral.com/mt/archives/2007/08/light_therapy_a.html